CLINICAL TRIAL: NCT00024037
Title: A Phase II/III Blinded Randomized Trial to Determine the Efficacy of Low Energy Diode Laser Therapy (650 nm or 780 nm) to Prevent Oral Mucositis Following Bone Marrow Transplantation
Brief Title: Laser Therapy in Preventing Oral Mucositis in Patients Undergoing Bone Marrow Transplantation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: 1001.00; FHCRC-1001.00; NCI-G01-2008; CDR0000068886 (Registry Identifier: PDQ); NCT01005134 (obsolete NCT alias)
Record Dates: First submitted 2001-09-13; First posted 2004-02-27 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2010-06

CONDITIONS: Oral Complications
Keywords: oral complications

INTERVENTIONS:
Procedure: management of therapy complications

SUMMARY:
RATIONALE: Laser therapy may reduce the severity of symptoms and speed healing of oral mucositis. It is not yet known if laser therapy is effective in preventing oral mucositis.

PURPOSE: Randomized phase II/III trial to determine the effectiveness of laser therapy in preventing oral mucositis in patients who are undergoing bone marrow transplantation.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether low-energy laser therapy can prevent oral mucositis in patients undergoing bone marrow transplantation.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are randomized to one of three treatment arms. Arm I: Patients undergo low-energy laser therapy with visible red light (650 nm) daily over 15-20 minutes beginning on the first day of their transplant conditioning regimen and continuing until day 2 after bone marrow transplantation. Arm II: Patients undergo low-energy laser therapy with invisible infra-red light (780 nm) daily on the same schedule as in arm I. Arm III: Patients undergo sham laser therapy daily on the same schedule as in arm I. Patients are followed on days 3, 7, 10, 14, 18, 21, and 24.

PROJECTED ACCRUAL: A total of 66 patients (22 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: At risk of developing oral mucositis due to toxicity resulting from one of the following: Preparative chemoradiotherapy Multiple drug conditioning regimens Graft-versus-host disease (GVHD) prophylaxis

PATIENT CHARACTERISTICS: Age: Over 12 Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Able to carry out routine oral care No active oral, viral, bacterial, or fungal infections No active uncontrolled oral bleeding that would preclude laser therapy

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: Not currently enrolled on other protocols with oral mucositis as a stated end point (e.g., conditioning regimen toxicity trials or GVHD prophylaxis trials) No other concurrent investigational drugs or agents for the prevention or treatment of mucositis No concurrent photosensitizing agents

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-04; Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark M. Schubert, DDS, MSD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States